CLINICAL TRIAL: NCT03300830
Title: Molecular Characterization of Viral-associated Tumors, Tumors Occurring in the Setting of HIV or Other Immune Disorders and Castleman Disease
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170174; 17-C-0174
Record Dates: First submitted 2017-10-03; First posted 2017-10-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Human Immunodeficiency Virus; Castleman's Disease; Kaposi's Sarcoma; Viral-Associated Cancer
Keywords: Immunodeficiency; Viral-Associated Cancer; Kaposi Sarcoma Herpes Virus; Idiopathic Castleman Disease; Endogenous Retroviruses; Natural History
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Castleman Disease; Sarcoma, Kaposi; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: Viral-assoc. cancer; HIV-neg pts with cancer that occurs in HIV pos; KSHV-assoc. cancer or related diseases e.g. multicentric Castleman disease (MCD); retrovirus-induced cancer; Idiopathic Castleman disease

SUMMARY:
Background:

A person s genome is the collection of all their genes. A gene instructs individual cells to make proteins. Proteins are involved in all of our body s chemical processes. Genome sequencing allows researchers to find variations in genes. Some of these are normal and are not known to cause disease. Some variants are known to cause or affect diseases like cancer. Researchers want to study genetic variants in people with cancer who also have an immunologic disease like HIV.

Objective:

To study the biology of cancer in order to improve ways to prevent, detect, and treat it.

Eligibility:

Adults at least 18 years old with certain cancers and/or immunodeficiencies

Design:

Participants will be screened with medical history, physical exam, and lab tests.

Participants will give samples of one or more tissue type.

They may give blood or urine samples.

Researchers may get samples of tissue when participants have surgery or when the participants are on other protocols in the NCI.

Participants may have a procedure to have tissue samples removed.

Researchers may collect data from participant medical records.

Researchers will compare the genes in a participant s cancer tissue to their normal tissue. They may use the tissue cells to grow new cells in a lab.

Participants may be contacted about the results.

The samples will be stored for future research. No personal data will be kept with them.

...

DETAILED DESCRIPTION:
Background:

* The availability of high quality, clinically annotated patient samples is crucial for the study of biologic factors that influence the natural history of viral related malignancies, malignancies occurring in the setting of human immunodeficiency virus (HIV), and Castleman disease.
* Comprehensive genomic sequence of viral-associated malignancies, malignancies occurring in the setting of HIV, tumors hypothesized to be caused by endogenous retroviruses, and Castleman disease may identify diagnostic or prognostic disease signatures, and recurrent driver alterations that interact with viral factors, and may identify targets for new therapies.
* Comparison of transcriptomes and genomes between cancers or Castleman disease from HIV+ and HIV- individuals might identify novel non-human sequences that could potentially suggest the presence of transcripts from hitherto undiscovered oncogenic viral agents.

Objective:

-The primary objective of this protocol is to support molecular investigation of viral associated malignancies, malignancies occurring in the setting of HIV or other immunodeficiencies, and Castleman disease, by accrual of high quality, clinically annotated tissue from such participants as well as participants with tumors that may serve as appropriate controls.

Eligibility:

* Age >=18 years
* HIV or other acquired immunodeficiency and cancer or
* Viral-associated cancer or
* HIV-negative with cancer that commonly occurs in people with HIV or
* Kaposi sarcoma herpes virus (KSHV)-associated malignancy or related diseases, such as Multicentric Castleman Disease (MCD) or
* Idiopathic Castleman disease or
* Tumors that are hypothesized to be caused by endogenous retroviruses

Design:

* Samples will be processed using project specific collection and processing protocols.
* Collection of non-tumor specimens will generally be performed to obtain germ-line genetic material. The results between tumor and normal DNA will be analyzed to identify the somatic changes present in the cancer tissues.
* Alterations to be evaluated may include: detection of chromosomal changes, such as, but not limited to, amplification, deletions, loss of heterozygosity, translocations, etc.; as well as expression profiling and detection of transcripts resulting from translocations and mutations, including single nucleotide variants, insertions, deletions, etc.
* Multiple forms of project specific analyses may be performed, including evaluation of polymorphisms, mutations, gene expression, circulatory and tissue-based biomarkers, whole exome sequencing, and clinical pathologic correlation based on project specific statistical and bioinformatics plans.
* Alterations may also be analyzed within the context of biological pathways and systems biology being evaluated in a given project.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants with one or more of the following:

* HIV or other acquired immunodeficiency and cancer
* Viral-associated cancer or cancer hypothesized to be caused by a virus
* HIV-negative participants with cancer that commonly occurs in people with HIV

  --KSHV-associated malignancy or related diseases, such as Multicentric Castleman Disease (MCD)
* A malignancy hypothesized to be caused by an endogenous retrovirus
* Idiopathic Castleman disease

Cancer diagnoses will be confirmed by the NCI Laboratory of Pathology (LP). A biopsy will be collected if sufficient archival tissue is not available.

* Age >=18 years.
* ECOG performance status <=2 (Karnofsky >=60%) if biopsy to be performed is solely for the purposes of this protocol. Any ECOG performance status will be allowed if biopsy required for participant care or another NIH protocol that allows lower performance status or if enrollment on this protocol is only for the purposes of studying tissue that has already been collected.
* Participants must have signed or be willing to sign an IRB-approved informed consent document that permits the use of the tumor and other samples for genomic-based molecular characterization projects. Telephone consent for use of archival tissue or tissue collected on another protocol or standard participant care will be permitted.
* Co-enrollment on other HAMB, NCI, or NIH protocols is allowed

EXCLUSION CRITERIA:

* Inability to provide informed consent.
* Pregnancy: Pregnant women will not be allowed to participate in this study because there is not a potential benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be participants referred by HIV providers and those who provide primary care to the African immigrant community.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2037-06-07 (Estimated); Study Completion 2037-06-25 (Estimated)

PRIMARY OUTCOMES:
Tissue collection | Time of collection
  Molecular data from viral associated malignancies, malignancies occurring in the setting of HIV or other immunodeficiencies, and Castleman disease

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians

REFERENCES:
- [Derived] Ramaswami R, Tagawa T, Mahesh G, Serquina A, Koparde V, Lurain K, Dremel S, Li X, Mungale A, Beran A, Ohler ZW, Bassel L, Warner A, Mangusan R, Widell A, Ekwede I, Krug LT, Uldrick TS, Yarchoan R, Ziegelbauer JM. Transcriptional landscape of Kaposi sarcoma tumors identifies unique immunologic signatures and key determinants of angiogenesis. J Transl Med. 2023 Sep 22;21(1):653. doi: 10.1186/s12967-023-04517-5. PMID 37740179
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0174.html